CLINICAL TRIAL: NCT06106139
Title: The Effectiveness of Ketogenic Diet in Preventing or Improving Thrombocytopenia in Cancer Patients Undergoing Chemotherapy: a Randomized Controlled Single Blind Study
Brief Title: Ketogenic Diet Improves Thrombocytopenia in Cancer Patients
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baoling Guo (Other)
Responsible Party: Sponsor-Investigator, Baoling Guo, associate chief physician, Fujian Medical University
Organization: Fujian Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LYSY20230510
Record Dates: First submitted 2023-06-01; First posted 2023-10-30 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Ketogenic Diet

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normal diet group (No Intervention): This group of patients follows the "Dietary Guidelines for Chinese Residents (2022)" to ensure balanced nutrition, with daily calorie intake ranging from 1600 to 2400 kcal.
- Strict ketogenic diet group (Experimental): the patients ate ketogenic biscuits or ketogenic foods provided by the researchers every day. During the study, the patients were not allowed to drink any drinks or eat other foods except drinking water, so as to ensure that the daily intake of calories was roughly the same as that of the normal diet group.
  Interventions: Dietary Supplement: Strict ketogenic diet group
- Cyclic ketogenic diet group (Experimental): the patients took 7 days as a cycle, and 7 days of strict ketogenic diet+7 days of normal diet as a cycle. During the strict ketogenic diet, the patient should eat the ketogenic biscuit or ketogenic food provided by the researcher every day, and should not drink any beverage or eat other food except drinking water; During the normal diet period, patients followed the "Dietary Guidelines for Chinese Residents (2022)" to ensure nutritional balance. During the study period, patients were guaranteed to eat approximately the same amount of calories per day as the normal diet group.
  Interventions: Dietary Supplement: Cyclic ketogenic diet group
- Autonomous ketogenesis group (Experimental): Patients choose ingredients for cooking and consumption under the guidance of researchers, ensuring that the nutritional composition is about 90% fat, 10% protein, and can contain a small amount of carbohydrates (10%). The daily calorie intake is around 1600~2400 kcal.
  Interventions: Dietary Supplement: Autonomous ketogenesis group

INTERVENTIONS:
Dietary Supplement: Strict ketogenic diet group — the patients ate ketogenic biscuits or ketogenic foods provided by the researchers every day. During the study, the patients were not allowed to drink any drinks or eat other foods except drinking water, so as to ensure that the daily intake of calories was roughly the same as that of the normal diet group.
  Arms: Strict ketogenic diet group
Dietary Supplement: Cyclic ketogenic diet group — the patients took 7 days as a cycle, and 7 days of strict ketogenic diet+7 days of normal diet as a cycle. During the strict ketogenic diet, the patient should eat the ketogenic biscuit or ketogenic food provided by the researcher every day, and should not drink any beverage or eat other food except drinking water; During the normal diet period, patients followed the "Dietary Guidelines for Chinese Residents (2022)" to ensure nutritional balance. During the study period, patients were guaranteed to eat approximately the same amount of calories per day as the normal diet group.
  Arms: Cyclic ketogenic diet group
Dietary Supplement: Autonomous ketogenesis group — Patients choose ingredients for cooking and consumption under the guidance of researchers, ensuring that the nutritional composition is about 90% fat, 10% protein, and can contain a small amount of carbohydrates (10%). The daily calorie intake is around 1600~2400 kcal.
  Arms: Autonomous ketogenesis group

SUMMARY:
The main purpose of this study is to evaluate whether dietary intervention through ketogenic diet can prevent or improve chemotherapy related thrombocytopenia in cancer patients.

DETAILED DESCRIPTION:
In the study, 80 patients with malignant solid tumors undergoing chemotherapy were randomly assigned to the normal diet group, the strict ketogenic diet group, the circulating ketogenic diet group, and the autonomous ketogenic group. During the chemotherapy period, the corresponding dietary intervention was carried out, and the clinical data of patients before and after treatment were collected, including blood routine, blood ketone concentration, weight, blood sugar, blood lipids, adverse events, and changes in platelets before and after chemotherapy, Statistical analysis of data such as the change degree of platelets and the incidence of adverse events in each diet group before and after treatment was carried out to evaluate the impact of ketogenic diet on clinical indicators and adverse reactions of chemotherapy in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 90, regardless of gender
* ECOG score ≤ 2 points
* Received or expected to receive radiotherapy and chemotherapy during tumor activity
* Body mass index 19-29
* Conscious and autonomous eaters

Exclusion Criteria:

* Patients with basic diseases of diabetes
* Complications such as severe liver and kidney dysfunction or digestive tract obstruction, inability to eat
* Those who have a preference for food and have strict requirements for dietary taste
* Disagree to sign informed consent
* Those whose physical conditions are determined by the doctor to be impermissible

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-05-12 (Estimated); Primary Completion 2024-06-10 (Estimated); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
thrombocytopenia | During radiotherapy and chemotherapy, approximately 3 months